CLINICAL TRIAL: NCT01698541
Title: Generic Tacrolimus in the Elderly - Prograf® vs Tacni®
Acronym: GenTac
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anders Åsberg, Professor, University of Oslo School of Pharmacy
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GenTac-12; NCT01798758 (obsolete NCT alias)
Record Dates: First submitted 2012-09-21; First posted 2012-10-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: End Stage Renal Disease
Keywords: Renal; Transplantation; Elderly
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacni (Experimental): Tacrolimus administered as generic formulation Tacni in accordance with standard protocol at the transplant center
  Interventions: Drug: Tacrolimus
- Prograf (Active Comparator): Tacrolimus administered as Prograf in according to standard protocol at the transplant center
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tested generic
  Other Names: Tacrolimus formualted as the generic Tacni
Drug: Tacrolimus — Original formulation used as comparator
  Other Names: Tacrolimus formualted as the original Prograf

SUMMARY:
Test bioequivalence of generic tacrolimus (Tacni), using original tacrolimus (Prograf) as comparator, in elderly (>60 yr) renal transplant recipients

DETAILED DESCRIPTION:
12-hour pharmacokinetic investigations performed on each formulation in each patient at steady-state. Patients will be randomized with regards to which formulation to start with. 1-2 weeks between each PK investigation.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients that will receive Tac as part of their immunosuppressive therapy.
* Recipients 60 years of age or older.
* Signed informed consent.

Exclusion Criteria:

* Diabetes mellitus (WHO criteria).
* Concomitant treatment with: diltiazem, verapamil, phenytoin, carbamazepin, fluconazole, ketoconazole, voriconazole, erythromycin, clarithromycin.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | 10 weeks
  Bioequivalence will be assessed at steady-state by comparing both AUC(0-12) and Cmax ratios for generic:original-ratios and applying the stricter 90-111% bioequivalence criteria.
  AUC(0-12) will be assessed by trapezoidal rule and Cmax will be the highest actually measured concentration.

SECONDARY OUTCOMES:
Population model validation | 10 weeks
  Use these new patient data to verify previously developed population pharmacokinetic model for tacrolimus.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, PhD, Study Chair — University of Oslo
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway